CLINICAL TRIAL: NCT01172327
Title: Evaluation of a Self-directed, Packaged Physical Activity Program for Adults With Arthritis
Brief Title: Self-Directed Exercise Program for Adults With Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Sara Wilcox, Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00004658
Record Dates: First submitted 2010-05-17; First posted 2010-07-29 (Estimated); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Arthritis; Osteoarthritis; Rheumatoid Arthritis; Fibromyalgia
MeSH Terms: conditions — Arthritis; Osteoarthritis; Arthritis, Rheumatoid; Fibromyalgia | interventions — Nutritional Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Multicomponent exercise (Experimental): This arm is a self-directed, multicomponent, exercise intervention. Participants exercise on their own and follow a progressive stepped program that occurs in the following order: cardiorespiratory exercises, flexibility exercises, strength (upper and lower body) exercises, and balance exercises. Participants also complete a daily log of their exercises and return the logs every week for 12 weeks.
  Interventions: Behavioral: Multicomponent exercise
- Nutrition (Active Comparator): This arm is a self-directed nutrition intervention. Participants follow a progressive stepped program that occurs in the following order: fruits, vegetables, grains, meat and beans. Participants also complete a daily log of their dietary intake and return the logs every week for 12 weeks.
  Interventions: Behavioral: Nutrition

INTERVENTIONS:
Behavioral: Multicomponent exercise — This intervention is a self-directed, multicomponent, exercise intervention. Participants exercise on their own and follow a progressive stepped program that occurs in the following order: cardiorespiratory exercises, flexibility exercises, strength (upper and lower body) exercises, and balance exercises. Participants also complete a daily log of their exercises and return the logs every week for 12 weeks. The active intervention phase is 12 weeks.
  Arms: Multicomponent exercise
Behavioral: Nutrition — This arm is a self-directed nutrition intervention. Participants follow a progressive stepped program that occurs in the following order: fruits, vegetables, grains, meat and beans. Participants also complete a daily log of their dietary intake and return the logs every week for 12 weeks. The active intervention lasts for 12 weeks.
  Arms: Nutrition

SUMMARY:
The purpose of this study is to examine the effectiveness and safety of a self-directed physical activity program relative to a self-directed dietary program in adults with arthritis. A process evaluation will also be conducted to examine program reach, participation/dose, fidelity, and participant compatibility/satisfaction.

DETAILED DESCRIPTION:
Physical activity is a critical component of arthritis disease management. It also reduces the risk for other chronic comorbid conditions in people with arthritis. Yet, most adults with arthritis are not sufficiently active at the level needed to achieve benefits. Existing group-based arthritis exercise programs reach only a very small percentage of the population. The overall purpose of this study is to test a self-directed and low-cost multicomponent physical activity program for people with arthritis on outcomes including symptoms of arthritis, lower body strength, functional aerobic capacity, flexibility, physical activity, arthritis self-efficacy and disability, upper body strength, balance, gait, and depressive symptoms. The second primary aim is to evaluate the safety of the physical activity program. The third primary aim is to conduct a process evaluation to examine program reach, participation/dose, fidelity, and participant compatibility/satisfaction. Adults aged 18 years and older with arthritis will be recruited from the midlands area of South Carolina. After completion of a baseline visit, participants will be randomized in equal numbers to the 12-week physical activity program (First Step to Active Health®) or the 12-week attention-control group (Steps to Healthy Eating). The attention control intervention will have the same "look and feel" as the physical activity intervention and will require similar activities such as self-monitoring of behavior. Follow-up measurements will take place post-program (12-weeks) and 6 months post-program (i.e., 9 months post-randomization). If First Step to Active Health® is shown to be effective, it could be widely disseminated for a very low cost, thus having the potential to make a tremendous public health impact on the burden of arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported, health care provider-diagnosed arthritis (CDC definition)
* 18+ years of age
* Self-reported symptoms of joint pain, stiffness, tenderness, decreased range of motion, redness and warmth, deformity, crackling or grating, or fatigue
* Able to read and write in English

Exclusion Criteria:

* Another member of household is participating in study
* Plans to move from the Columbia, SC area in the next 9 months
* Unable to walk longer than 3 minutes without taking a rest
* Unable to stand without assistance for more than 2 minutes
* Cannot sit in a chair without arms for more than 5 minutes
* Measured resting blood pressure >160/100
* Positive response to PAR-Q question(s)
* Had a fall in the past year that required medical assistance
* Pregnant or breastfeeding
* Uses insulin to manage diabetes
* Participating in another research study that includes an intervention or drug
* Participates in 3+ days of structured moderate-intensity exercise for 30+ minutes per day
* Participates in 2+ days of strength building exercises for 20+ minutes per day

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 401 (Actual)
Dates: Start 2009-09; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Symptoms of arthritis | 12 weeks
  Visual numeric scales to assess pain, fatigue, and stiffness
Lower body strength | 12 weeks
  The 30-second chair stand will assess lower body strength.
Functional exercise capacity | 12 weeks
  The six-minute walk will assess functional exercise capacity
Flexibility | 12 weeks
  The sit-and-reach test will assess flexibility
Physical activity | 12 weeks
  The Community Health Activities Model Program for Seniors Physical Activity (CHAMPS) Questionnaire will assess physical activity participation
Arthritis management self-efficacy | 12 weeks
  The Arthritis Self-Efficacy Scale will assess confidence in managing arthritis symptoms

SECONDARY OUTCOMES:
Disability | 12 weeks
  The Health Assessment Questionnaire (HAQ) will assess disability
Upper body strength | 12 weeks
  The grip strength test (kg/lbs of force) will assess upper body strength
Balance | 12 weeks
  Postural sway will be measured with the AMTI force platform to determine COP displacement, COP velocity, and 95th eclipse
Gait | 12 weeks
  GAITRite will assess components of gait including cadence, step time, cycle time, step length, stride length, and velocity
Depressive symptoms | 12 weeks
  The short form of the Center for Epidemiological Studies Depression scale (CES-D) will assess depressive symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Sara Wilcox, PhD, Principal Investigator — University of South Carolina
Locations (1):
- University of South Carolina Prevention Research Center, Columbia, South Carolina, United States

REFERENCES:
- [Derived] Baruth M, Wilcox S, Jake-Schoffman DE, Schlaff RA, Goldufsky TM. Effects of a Self-Directed Nutrition Intervention Among Adults With Chronic Health Conditions. Health Educ Behav. 2018 Feb;45(1):61-67. doi: 10.1177/1090198117709317. Epub 2017 Jun 3. PMID 28580795
- [Derived] Wilcox S, McClenaghan B, Sharpe PA, Baruth M, Hootman JM, Leith K, Dowda M. The steps to health randomized trial for arthritis: a self-directed exercise versus nutrition control program. Am J Prev Med. 2015 Jan;48(1):1-12. doi: 10.1016/j.amepre.2014.08.006. Epub 2014 Nov 6. PMID 25441237
- [Derived] Schoffman DE, Wilcox S, Baruth M. Association of body mass index with physical function and health-related quality of life in adults with arthritis. Arthritis. 2013;2013:190868. doi: 10.1155/2013/190868. Epub 2013 Dec 12. PMID 24392226